CLINICAL TRIAL: NCT03684447
Title: Neural and Antidepressant Effects of Propofol
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, Principal Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00116093
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Participants randomized to the high dose will exit the study after treatment. Participants randomized to the low dose who have not experienced response are able to crossover to the high dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol High Dose (Experimental): high propofol injectable, individually dosed, three times per week
  Interventions: Drug: Propofol
- Propofol Low Dose (Experimental): low propofol injectable, individually dosed, three times per week
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Series of 6 treatments with propofol.
  Other Names: Diprivan
  Arms: Propofol High Dose
Drug: Propofol — Series of 6 treatments with propofol. May be able to cross over and receive 6 additional treatments with the high dose of propofol.
  Other Names: Diprivan
  Arms: Propofol Low Dose

SUMMARY:
This study will compare the antidepressant effects of propofol at two different doses while measuring potential treatment-related biomarkers.

DETAILED DESCRIPTION:
Aim 1: Compare the clinical antidepressant effects of high-dose versus low-dose propofol.

Aim 2: Characterize the dose-dependent effects of propofol on brain function and gene expression

ELIGIBILITY:
Inclusion Criteria:

Age 18-55 years Diagnosis of major depressive disorder or bipolar disorder Current moderate-to-severe depressive episode Episode duration more than 2 months and less than 5 years Failure of at least 2 adequate antidepressant medication trials within the past 2 years 16-item Quick Inventory of Depressive Symptomatology, self-rated (QIDS) > 10 24-item Hamilton Depression Rating Scale (HDRS) > 18

Exclusion Criteria:

Contraindication to propofol, egg lecithin, soybean oil, or other study drugs Lifetime history of a serious suicide attempt(Gvion and Levi-Belz, 2018) Recent suicidal behavior(past 3 months) Body mass index > 40 kg/m2 Daily use of benzodiazepine, opioid, ACE inhibitor, or ARB medication Symptomatic coronary artery disease or heart failure Poorly controlled hypertension or diabetes Abnormal kidney or liver function Pregnant or breast feeding Traumatic brain injury or significant neurologic signs (past year) Substance use disorder, moderate-to-severe(past 3 months) Obsessive compulsive disorder (past month) Post-traumatic stress disorder (past month) Schizophrenia-spectrum disorder (lifetime) Neurocognitive disorder (past year) Personality disorder as a current focus of treatment ECT within the past 3months Inappropriate for ECT, or poor response to ECT within the past 5 years Incompetent to provide consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | approximately 17 days after randomization
  24-item Hamilton Depression Rating Scale, total score Higher values represent more severe depressive symptoms Maximum score, 76; minimum score, 0 Remission defined as total score < 10 Response defined as decrease of total score from baseline of 50% or greater

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | approximately 36 days after randomization
  24-item Hamilton Depression Rating Scale, total score Higher values represent more severe depressive symptoms Maximum score, 76; minimum score, 0 Remission defined as total score < 10 Response defined as decrease of total score from baseline of 50% or greater

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Mickey, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University Neuropsychiatric Institute, Salt Lake City, Utah, United States